CLINICAL TRIAL: NCT04990765
Title: Virtual Reality-Assisted Cognitive Behavioral Therapy for Alcohol Dependence: A Pilot Study (CRAVR-Pilot)
Brief Title: Virtual Reality-Assisted Cognitive Behavioral Therapy for Alcohol Dependence (CRAVR-Pilot)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Psychiatric Centre Rigshospitalet (Other)
Collaborators: The Novavì outpatient clinics, Copenhagen (Unknown)
Responsible Party: Principal Investigator, Anders Fink-Jensen, MD, DMSci, Professor, MD, DMSci, Psychiatric Centre Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRAVRPILOT
Record Dates: First submitted 2021-06-15; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Alcohol Dependence, in Remission; Addiction, Alcohol
Keywords: Alcohol; Addiction; Virtual Reality; Exposure Therapy; Cognitive Behavioral Therapy
MeSH Terms: conditions — Alcoholism; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: single-blinded, randomized, controlled
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Cognitive Behavioral Therapy (VRCBT) (Experimental): The VR exposure is performed to induce alcohol craving during the therapy session, in order to trigger a lifelike response to alcohol, while the therapist is present and able to train the participant in applying CBT-based coping strategies to deal with the alcohol cravings.
  Interventions: Behavioral: Virtual Reality Cognitive Behavioral Therapy (CRAVR)
- Cognitive Behavioral Therapy (CBT) (Active Comparator): CBT is made up of the following elements: i) recognition (ii) avoiding and (iii) overcoming drinking cravings in high-risk situations with the aim of preventing relapse.
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: Virtual Reality Cognitive Behavioral Therapy (CRAVR) — Participants in the intervention group will scheduled for 3 weekly treatment sessions based on manualized cognitive behavioral therapy assisted with alcohol-related high risk situations (6 different scenes from a restaurant) in virtual reality. From scene 1 to scene 6, alchol-related cues increase in intensity in order to perform gradual exposure therapy as a part of CBT. Furthermore, VR scenes are used in CBT to induce craving for coping strategy skill training and cognitive analysis.
  Arms: Virtual Reality Cognitive Behavioral Therapy (VRCBT)
Behavioral: CBT — The active comparator receives 3 conventional cognitive behavioral therapy sessions with 1 week intervals.
  Arms: Cognitive Behavioral Therapy (CBT)

SUMMARY:
The pilot study is a single-blinded, randomized, controlled, 2 months clinical trial. The objective is to investigate the feasibility, effects and side-effects of virtual reality-assisted cognitive behavioral therapy (VR-CBT) vs. cognitive behavioral therapy (CBT) on alcohol intake in patients with a diagnosis of alcohol dependence.

DETAILED DESCRIPTION:
Pilot study rational:

Prior to the major randomized clinical trial, a total of 10 participants with alcohol dependence are included in a pilot trial. This is done to examine the feasibility of the following elements:

i) adherence to the intervention and drop-outs ii) the therapists' theoretical and practical abilities to use the virtual reality (VR) equipment iii) the time spent on virtual reality during the therapy session iv) the need for technical support v) the collaboration in the project group and vi) the participants' experience of virtual reality-assisted cognitive behavioral therapy (VRCBT).

During the pilot trial, patients receive standardized alcohol treatment for alcohol dependence at the Novavis outpatient clinics based on national guidelines from health authorities. Three of the therapy sessions contain VR-CBT.

Recruitment of participants:

Patients seeking alcohol treatment in the Novaví outpatient clinics are informed orally and in writing about the research project, and if they are interested, an information meeting is booked. If patients exhibit abstinence, these are treated prior to a possible information meeting by doctors and nurses in Novaví. If the patient wishes to participate and meets the inclusion criteria, informed consent is obtained, and screening is conducted using questionnaires described below.

Screening:

At the screening sessions, patiens medical history is obtained, as well as patients' alcohol intake over the past 30 days is recorded via Timeline Follow-back (TLFB). Patients are also asked about previous alcohol dependence treatment and general information about psychosocial factors incl. education, work, marital status, and functional level using Global Assessment of functioning (GAF). In addition, alcohol-related problems are assessed using the Alcohol Users Identification Test (AUDIT), abstinence using the Clinical Institute Withdrawal Assessment of Alcohol Scale Revised (CIWA-Ar), intake of other drugs using the Drug User Identification Test (DUDIT), alcohol craving using the Penn Alcohol Craving Scale (PACS). The Becks questionnaires, Depression Inventory 2 (BDI-II) and Beck's Anxiety Inventory (BAI), are included to assess the degree of anxiety and depression, and in addition, tests of mental function are performed using the Screening for Cognitive Impairment in Psychiatry (SCIP).

Intervention:

Included participants will in collaboration with their therapist schedule a standard course of treatment based on national guidelines from health authorities. After inclusion, participants are randomized to either:

1. 3 sessions of VR-CBT (Group A)
2. CBT without VR (Group B, control group)

The participants in group A are exposed to VR-simulated high-risk situations filmed in a restaurant to trigger alcohol cravings of which the participants are subsequently trained to handle by trained therapists using CBT-based techniques.

The participants in group B receive the same treatment without VR exposure. There will be weekly therapy sessions of approx. 1 hour for 3 weeks.

The intervention deviates from standard treatment, as none of the participants receive pharmaceutical alcohol treatment during the treatment period except for abstinence treatment if needed.

Randomization and blinding:

After screening the patient (ensuring that all inclusion criteria and no exclusion criteria are met) the patient is included. Participants are randomly allocated to either VR-CBT og CBT, 5 participants in each group. After randomization, the therapist ensures that the participant receives the correct treatment and performs the alcohol craving assessment during each VR-CBT session unblinded using visual analog score (VAS). The study staff conducting the remaining data collections and the entire data analysis are blinded, until the database is opened at the end of the study.

Follow-up:

Each patient must attend a follow-up visit 1 week and 1 month after the last session (session 3), where data collection will take place using the before mentioned questionnaires. The follow-up visit will be approx. 1 hour.

Statistical analysis:

All statistical analyzes are performed using the intention-to-treat principle, where all patients who have become randomized and has received a minimum of 1 session of VRCBT (group A) or CBT without VR (group B), is included in the analysis. Missing data are implemented through the multiple imputation method and the analyzes are performed in the program "R" with alpha = 0.05 and 2-sided test. All continuous effect measures are analyzed using ANOVA from baseline to most recent measurement, and categorical data are analyzed using chi2 analysis. All data distributions will be assessed for normality by visual inspection of histogram and by Q-Q plots. If data is not normally distributed, log transformation is performed, and if this is not successful, non-parametric testing is used.

ELIGIBILITY:
Inclusion Criteria:

* Informed oral and written consent
* Meets criteria for alcohol dependence syndrome according to International Classification of Diseases (ICD) 10, WHO & Diagnostic and Statistical Manual of Mental Disorder (DSM-5)
* Age 18 - 70 years old (both included)
* Minimum 5 'heavy drinking days' in the last month, which is defined as an alcohol intake above 60/48 grams or 5/4 items per. day for resp. men and women over the past 30 days

Exclusion Criteria:

* Other active substance use defined by DUDIT score> 6 (for men)> 2 (for women) and meet the criteria for other drug dependence according to ICD-10 (excluding nicotine)
* Does not speak or understand Danish
* Mental retardation or known severe psychiatric illness or other condition where it is assessed that will interfere with participation eg severely impaired vision or hearing.
* Medical alcohol treatment (disulfiram, acamprosate, naltrexone or nalmefen) within the latest 4 weeks and during the treatment period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-10-20 (Estimated); Study Completion 2021-10-20 (Estimated)

PRIMARY OUTCOMES:
Reduction in total alcohol consumption | From baseline to 1 week and 1 month after the third and final treatment session
  Percent reduction in alcohol consumption, defined as "x" grams of alcohol for past 30 days. This will be registered using the Timeline-Follow-Back (TLFB) method.

SECONDARY OUTCOMES:
Reduction in heavy drinking days | Baseline,1 week and 1 month follow-up
  Based on the past 30 days of alcohol consumption using time line follow-back (TLFB), heavy drinking days are evaluated. 1 heavy drinking day consists of alcohol consumption exceeding 60/48 grams for men and women respectively.
Reduction in Alcohol Users Identification Test (AUDIT) score | Baseline, 1 week and 1 month follow-up
  Screening for excessive drinking. Higher score = worse outcome
Reduction in Drug User Identification Test (DUDIT) score | Baseline, 1 week and 1 month follow-up
  Identification of individuals with drug-related problems. Higher score = worse outcome
Reduction in Penn Alcohol Craving Scale (PACS) score | Baseline, 1 week and 1 month follow-up
  Assessing alcohol craving. Higher score = worse outcome
Screening for Cognitive Impairment in Psychiatry (SCIP) score | Baseline, 1 week and 1 month follow-up
  The 20 minute test is a scale developed for screening cognitive deficits. Higher score = better outcome
Reduction in Global Assessment of functioning (GAF) score | Baseline, 1 week and 1 month follow-up
  GAF measures to what degree a person's symptoms affect their daily functioning on a scale of 0 to 100. Higher score = better outcome
Becks Anxiety Inventory (BAI) score | For baseline to 1 week and 1 month follow-up
  Measures the severity of anxiety. Higher score = worse outcome
Becks Depression Inventory 2 (BDI-II) score | For baseline to 1 week and 1 month follow-up
  Measures the severity of depression. Higher score = worse outcome
Simulator Sickness Questionnaire (SSQ) | Evaluated in each session
  Measures whether participants experience symptoms of simulator sickness while in Virtual Reality. Higher score = worse outcome
VR-induced craving on a visual analog scale (VAS) | Evaluated in each session
  For each of the 6 VR-scenes, craving is evaluated before, during and after exposure.
VR-induced thoughts, emotions, physiological reactions and behavior | Evaluated in each session

CONTACTS AND LOCATIONS:
Locations (1):
- Novavi ambulatorierne, Copenhagen, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thaysen-Petersen D, Hammerum SK, Vissing AC, Oestrich IH, Nordentoft M, During SW, Fink-Jensen A. Virtual reality-assisted cognitive behavioral therapy for patients with alcohol use disorder: a randomized feasibility study. Front Psychiatry. 2024 Feb 14;15:1337898. doi: 10.3389/fpsyt.2024.1337898. eCollection 2024. PMID 38419905